CLINICAL TRIAL: NCT01294358
Title: Regional Chemotherapy in Locally Advanced Pancreatic Cancer: RECLAP Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udo Rudloff, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110099; 11-C-0099; P10764 (Other: National Institutes of Health Clinical Center (CC))
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Histologically or Cytologically Confirmed Pancreatic Ca; Unresectable or Borderline Resectable Pancreatic Ca
Keywords: Pancreatic Cancer; Regional Therapy; Selective Arterial Infusion; Locally Advanced Disease
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine Dose Escalation (Experimental): gemcitabine dose escalation
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
  Other Names: Gemzar

SUMMARY:
Background:

- Pancreatic cancer is difficult to treat because by the time most cases are diagnosed, the tumors are too large to be removed surgically. Standard intravenous chemotherapy may shrink some of the tumor, but even with chemotherapy only about 25 percent of patients will live for 1 year following diagnosis. Several preliminary studies have shown that it is safe to give chemotherapy directly into the pancreas in the area of the tumor, and that giving gemcitabine over a longer period increases the amount of drug that is available to the tumor. Researchers are interested in studying whether giving the approved pancreatic cancer chemotherapy drug gemcitabine directly into the pancreas in the area of the cancer and at a slow rate of infusion is a safe and effective treatment.

Objectives:

- To test the safety and effectiveness of administering gemcitabine directly to a pancreatic tumor at a slow rate of infusion.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with pancreatic cancer that is currently too large to be removed surgically but has not yet spread to other organs.

Design:

* Participants will be screened with a full medical history and physical examination, blood and urine tests, and imaging studies.
* Participants will undergo pancreatic angiography and embolization, during which a catheter will be threaded into the blood vessels near the pancreas and a contrast dye will be used to show the blood vessels supplying the tumor. These blood vessels will then be surgically closed off.
* After the embolization, gemcitabine will be given as an infusion into the area around the tumor over 24 hours.
* Participants will return to the clinical center every 2 weeks after the first infusion for additional infusions of gemcitabine, using the same procedures as above. Participants will be monitored with frequent blood tests and imaging studies.
* Two weeks after the fourth treatment (course 1), participants will have more imaging studies, a physical examination, and blood tests. If the tumor is shrinking, participants will have two more courses of treatment (eight more infusions of gemcitabine).
* Participants will have followup visits every 3 months for 2 years following the last treatment and then every 6 months.

DETAILED DESCRIPTION:
Background:

* Pancreatic cancer is the fourth leading cause of cancer death in the United States.
* Surgery offers the only chance at cure; however, less than 20% of patients are considered resectable at initial presentation.
* A common reason for being classified as unresectable is loco-regional advanced disease.
* Several phase I studies of regional administration of chemotherapy have proven safe.
* The main advantage of pancreatic cancer targeted arterial perfusion of Gemcitabine is achievement of higher local bio-available active drug levels at the tumor bed.
* The Regional Chemotherapy in Locally Advanced Pancreatic Cancer (RECLAP) trial is a phase I trial offering highly selective 24-hour intra-arterial administration of Gemcitabine via a subcutaneous port for patients with unresectable locally-advanced pancreatic cancer.

Objectives:

Primary Objective:

* To evaluate feasibility and toxicity of intra-arterial gemcitabine therapy (dose limiting toxicity (DLT)).
* To establish the maximum tolerated dose (MTD)

Secondary Objectives:

* To evaluate response rate using Response Evaluation Criteria in Solid Tumors (RECIST), positron emission tomography (PET), magnetic resonance imaging (MRI) and computed tomography (CT) perfusion criteria (European Association for the Study of the Liver (EASL))
* To determine progression free and overall survival.
* To evaluate the conversion rate from unresectable or borderline resectable to potentially resectable pancreatic cancer.
* To determine progression-free and overall survival.
* To analyze potential selection criteria to be used in future studies for patients who present with marginally unresectable or unresectable locally-advanced pancreatic cancer that might benefit from this approach.

Eligibility:

* Unresectable locally-advanced pancreatic cancer.
* 18 years old or greater with an Eastern Cooperative Oncology Group (ECOG) 0-2
* Laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to surgery or chemotherapy.
* No extra-pancreatic disease except regional lymph nodes.

Design:

* This is a dose escalation phase-I study.
* Patients considered unresectable due to locally-advanced pancreatic cancer will receive selective arterial perfusion of gemcitabine over 24 hours via a subcutaneous indwelling port.
* Treatment will be given on Days 1 and 14. One cycle = 4 weeks for up to six cycles.
* Three to six patients will be enrolled per dose cohort.
* 18 to 36 patients in 7 cohorts will be accrued plus 6 more patients at the maximum tolerated dose (MTD over 36 months. Patients will be evaluated every 2 cycles (8 weeks). Upon progression patients will be taken off study. If no progressive disease (PD), patients will continue up to 6 cycles.
* Chemotherapy na(SqrRoot) ve patients and patients who received previously chemotherapy including gemcitabine will be allowed, as this mode of administration has better bioavailability, offer potential for better biological effect and less systemic toxicity profiles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed locally advanced pancreatic adenocarcinoma or clinical and radiographic evidence of pancreatic cancer

Note: Patients with a limited disease burden outside the pancreas, who have undergone systemic chemotherapy for metastatic disease and have achieved a complete response on the metastatic lesions of greater than or equal to 6 months, and have no evidence of disease outside the pancreas at time of enrollment, are eligible.

* Disease must be evaluable
* Disease should be deemed unresectable by the MD Anderson criteria
* Patients may be chemo naive or have received prior chemotherapy (including Gemcitabine) and/or radiation
* Greater than or equal to 18 years of age
* Must be able to understand and sign the Informed Consent Document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) less than or equal to 2
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control during and for four months after receiving chemotherapy
* Hematology:

  * Absolute neutrophil count greater than 1300/mm(3) without the support of Filgrastim.
  * Platelet count greater than 75,000/mm(3).
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 3 times the upper limit of normal, unless patient carries a biliary stent. For these patients, to account for asymptomatic, transient elevations in transaminases ('transaminitis'), serum ALT/AST may be less than or equal to 5 times the upper limit of normal provided all other eligibility parameters are met.
  * Serum creatinine less than or equal to 1.8 mg/dl unless the measured creatinine clearance is greater than 60 mL/min/1.73 m(2)
  * Total bilirubin less than or equal to 2 mg/dl,
  * Prothrombin time (PT) within 2 seconds of the upper limit of normal or International Normalized Ratio (INR) less than or equal to 1.8
* No history of prior/other malignancies within the 2 years prior to enrollment with the exception of basal cell carcinoma

EXCLUSION CRITERIA:

* Metastatic disease including malignant ascites
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, heart failure
* Childs B or C cirrhosis or with evidence of severe portal hypertension by history, endoscopy, or radiologic studies
* Weight less than 40 kg
* Significant ascites, greater than 1000cc in the absence of peritoneal disease
* Concomitant medical problems that would place the patient at an unacceptable risk for the procedure
* Need for concurrent chemotherapy
* Discretion of the principal investigator (PI)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01-26 (Actual); Primary Completion 2014-07-23 (Actual); Study Completion 2014-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruix J, Sherman M, Llovet JM, Beaugrand M, Lencioni R, Burroughs AK, Christensen E, Pagliaro L, Colombo M, Rodes J; EASL Panel of Experts on HCC. Clinical management of hepatocellular carcinoma. Conclusions of the Barcelona-2000 EASL conference. European Association for the Study of the Liver. J Hepatol. 2001 Sep;35(3):421-30. doi: 10.1016/s0168-8278(01)00130-1. No abstract available. PMID 11592607
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Sener SF, Fremgen A, Menck HR, Winchester DP. Pancreatic cancer: a report of treatment and survival trends for 100,313 patients diagnosed from 1985-1995, using the National Cancer Database. J Am Coll Surg. 1999 Jul;189(1):1-7. doi: 10.1016/s1072-7515(99)00075-7. PMID 10401733
- [Derived] Davis JL, Pandalai P, Ripley RT, Langan RC, Steinberg SM, Walker M, Toomey MA, Levy E, Avital I. Regional chemotherapy in locally advanced pancreatic cancer: RECLAP trial. Trials. 2011 May 19;12:129. doi: 10.1186/1745-6215-12-129. PMID 21595953

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 patients were enrolled, but only 6 were treated. Patient # 7 was consented and registered but developed pancreatitis before treatment. This patient was not treated.
Groups:
- 18 mg/m(2)/24h: All participants that received at least one dose of gemcitabine 18 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
- 36 mg/m(2)/24h: All participants that received at least one dose of gemcitabine 36 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
- 72 mg/m(2)/24h: All participants that received at least one dose of gemcitabine 72 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
- 96 mg/m(2)/24h: All participants that received at least one dose of gemcitabine 96 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
- 115 mg/m(2)/24h.: All participants that received at least one dose of gemcitabine 115 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
Period: Cohort 1: 5/11/11-11/9/11
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h.
Started | 4 | 0 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: 6/9/11-9/17/12
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h.
Started | 0 | 6 (4 participants from 18mg move to 36mg and 2 additional participants were enrolled at this dose.) | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0
Not Completed | 0 | 2 | 0 | 0 | 0
Not completed — Disease progression | 0 | 2 | 0 | 0 | 0
Period: Cohort 3: 12/1/11-10/6/12
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h.
Started | 0 | 0 | 4 (4 participants from 36mg move to 72mg.) | 0 | 0
Completed | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0
Not completed — Disease progression | 0 | 0 | 2 | 0 | 0
Period: Cohort 4: 12/30/11-2/17/17
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h.
Started | 0 | 0 | 0 | 2 (2 participants from 72mg move to 96mg.) | 0
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — pt rec'd surgical resection of pancreas | 0 | 0 | 0 | 1 | 0
Period: Cohort 5: 3/8/12-3/9/12
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h.
Started | 0 | 0 | 0 | 0 | 1 (1 participant from 96mg move to 115mg.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — dose limiting toxicity grade 4 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants that received at least one dose of gemcitabine 18 mg/m(2)/24h, 36 mg/m(2)/24h, 72 mg/m(2)/24h, 96 mg/m(2)/24h, and/or 115 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.57 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Time from Diagnosis to Trial Enrollment [Median (Full Range); unit: Months] | 8.5 [5 to 16]
Serum CA 19-9 Level at the Time of Enrollment [Median (Full Range); unit: Units/ml] — The reference range of CA 19-9 is <37 units/mL.
  Units/ml | 133 [1.0 to 521.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT )
Description: Here is the number of participants with DLT. DLT is defined as follows: All grade 3 or greater toxicities with the exception of Grade 3 constitutional symptoms that persist for less than 72 hours, Grade 3 and 4 myelosuppression (neutrophils and thrombocytopenia) of less than 5 days duration. Grade 3 metabolic/laboratory events that are correctable within 24 hours. Events that are assessed by the principal investigator as clearly unrelated to the agent will not be considered DLTs (e.g., events directly related to catheter insertion, pain related to underlying disease).
Time Frame: Cycle 1 (4 weeks), for up to 6 cycles
Measure: Count of Participants; unit: Participants
Groups:
- 72 mg/m(2)/24h: All participants that received at least one dose of gemcitabine 72 mg/m(2)/24h
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
- 96 mg/m(2)/24h: All participants that received at least one dose of gemcitabine 96 mg/m(2)/24h
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 4 | 6 | 4 | 2 | 1
Participants | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: MTD (Maximum Tolerated Dose)
Description: The MTD is the highest dose that induces dose limiting toxicity (DLT) in no more than 2 patients among a cohort of 6 patients. If 1 or fewer patients experience dose limiting toxicity than the dose level will define the MTD. Only DLT's that occurred during cycle 1 of each dose level were used to determine the MTD.
Time Frame: Cycle 1 (4 weeks), for up to 6 cycles
Measure: Number; unit: mg/ml/24h
Groups:
- Gemcitabine Dose Escalation: All participants that received at least one dose of gemcitabine 18 mg/m(2)/24h, 36 mg/m(2)/24h, 72 mg/m(2)/24h, 96 mg/m(2)/24h, and/or 115 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
Arm/Group | Gemcitabine Dose Escalation
Number analyzed (Participants) | 6
mg/ml/24h | 115

3. Secondary Outcome: Response Using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Description: Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. Progression is at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or the appearance of one or more new lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum diameters while on study.
Time Frame: Every 2 cycles (8 weeks), up to 18 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 18 mg/m(2)/24h,: All participants that received at least one dose of gemcitabine 18 mg/m(2)/24h.
  gemcitabine dose escalation
  Gemcitabine: Gemcitabine starting dose was 18mg/m(2)/24h via infusion pump on days 1-14. One cycle = 4 weeks for up to six cycles. Three to six patients enrolled per dose cohort. Patients were dosed at successive higher doses until maximum tolerated dose or up to 165 mg/m(2)/24h.
Arm/Group | 18 mg/m(2)/24h, | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 4 | 6 | 4 | 2 | 1
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 0 | 0
  Stable disease | 4 | 4 | 2 | 2 | 0
  Progressive disease (PD) | 0 | 2 | 2 | 0 | 1

4. Secondary Outcome: Response Rate Using Positron Emission Tomography (PET)
Description: as for outcome 3
Time Frame: Every 2 cycles (8 weeks), up to 18 weeks
Population: Data was collected for this outcome measure but not analyzed because PET scans were inconsistently obtained. There was lack of scans pre-onstudy or while patient was on treatment. Without being able to make a pre-versus-on treatment comparison, this outcome measure was not done.
Arm/Group | Gemcitabine Dose Escalation | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Response Rate Using Magnetic Resonance Imaging (MRI)
Description: as for outcome 3
Time Frame: Every 2 cycles (8 weeks), up to 18 weeks
Population: This outcome measure was not done. No MRI data were collected. All patients had contrast-enhanced computed tomography (CTs,) and thus were followed for consistency reasons with CT and not MRI.
Arm/Group | Gemcitabine Dose Escalation | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Response Using Computed Tomography (CT) Perfusion Criteria European Association for the Study of the Liver (EASL1)
Description: as for outcome 3
Time Frame: Every 2 cycles (8 weeks), up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 4 | 6 | 4 | 2 | 1
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 0 | 0
  Progressive disease (PD) | 0 | 4 | 2 | 2 | 0
  Stable disease (SD) | 4 | 2 | 2 | 0 | 1

7. Secondary Outcome: Median Time to Progression
Description: Time to progression is the time between the first day of treatment to the day of disease progression. Progression is defined as at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or the appearance of one or more new lesions.
Time Frame: From first day of treatment to the day of progression, assessed up to 221 months
Measure: Median (Full Range); unit: Months
Arm/Group | Gemcitabine Dose Escalation
Number analyzed (Participants) | 6
Months | 2 [1 to 221]

8. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time between the first day of treatment to the day of death.
Time Frame: Overall survival was assessed through study completion, an average of 3 years.
Measure: Median (Full Range); unit: Months
Arm/Group | 18 mg/m(2)/24h, | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 4 | 6 | 4 | 2 | 1
Months | NA [NA to NA] — No deaths. | 9 [3 to 15] | 9 [3 to 16] | 15 [0 to 15] | NA [NA to NA] — No deaths.

9. Secondary Outcome: Number of Participants Who Converted From Unresectable or Borderline Resectable To Potentially Resectable Pancreatic Cancer
Description: Resectability is defined by the MD Anderson Resectability criteria: Resectable is no extension; normal fat plane between the tumor and the artery (superior mesenteric artery (SMA)). No extension (celiac axis/hepatic artery). Patent (superior mesenteric vein/portal vein (SMV/PV)). Borderline resectable is tumor abutment ≤180◦ (one half or less) of the circumference of the artery; periarterial stranding and tumor points of contact forming a convexity against the vessel improve chances of resection (SMA). Short-segment encasement/abutment of the common hepatic artery (typically at the gastroduodenal origin) (celiac axis/hepatic artery). Short-segment occlusion with suitable vessel above and below (SMV/PV). Locally advanced is encased (>180◦) (SMA). Encased and no technical option for reconstruction usually because of extension to the celiac axis/splenic/left gastric junction or the celiac origin (celiac axis/hepatic artery). Occluded and no technical option for reconstruction (SMV/PV).
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h. | 115 mg/m(2)/24h
Number analyzed (Participants) | 4 | 6 | 4 | 2 | 1
Participants | 0 | 0 | 0 | 1 | 1

10. Secondary Outcome: Number of Potential Selection Criteria to Be Used in Future Studies for Patients With Marginally Unresectable Or Unresectable Locally-Advanced Pancreatic Cancer
Description: Number of selection criteria that can be used for unresectable pancreatic cancer.
Time Frame: up to 2.5 years
Population: Data was not collected and this outcome measure was not done due to an insufficient number of participants enrolled in this study.
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned
Time Frame: Date treatment consent signed to date off study, approximately 2 years and 2 months and 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h | 115 mg/m(2)/24h
Number analyzed (Participants) | 4 | 6 | 4 | 2 | 1
Participants | 4 | 5 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately years, 2 months and 21 days.
Arm/Group | 18 mg/m(2)/24h | 36 mg/m(2)/24h | 72 mg/m(2)/24h | 96 mg/m(2)/24h. | 115 mg/m(2)/24h
All-Cause Mortality (participants affected / at risk) | 0/4 | 2/6 | 2/4 | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 0/4 | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 3/4 | 5/6 | 2/4 | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18 mg/m(2)/24h (N=4) | 36 mg/m(2)/24h (N=6) | 72 mg/m(2)/24h (N=4) | 96 mg/m(2)/24h. (N=2) | 115 mg/m(2)/24h (N=1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18 mg/m(2)/24h (N=4) | 36 mg/m(2)/24h (N=6) | 72 mg/m(2)/24h (N=4) | 96 mg/m(2)/24h. (N=2) | 115 mg/m(2)/24h (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 1 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, retained foreign body (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-11-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT01294358/Prot_000.pdf
  • Informed Consent Form (2012-11-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT01294358/ICF_001.pdf